CLINICAL TRIAL: NCT04234555
Title: What is the Nature of Pelvic Floor Muscle Involvement in Dyspareunia?
Status: Completed | Type: Observational
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Dr. Linda McLean, Professor in the School of Rehabilitation Sciences at the University of Ottawa., University of Ottawa
Other Study IDs: H-11-18-1183
Record Dates: First submitted 2020-01-10; First posted 2020-01-21 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Dyspareunia
Keywords: dyspareunia; electromyography; transcranial magnetic stimulation; pressure pain threshold; temporal summation; vaginismus; provoked vestibulodynia
MeSH Terms: conditions — Dyspareunia; Vaginismus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Provoked vestibulodynia (PVD): Provoked vestibulodynia (PVD) is characterized by severe sharp and/or burning pain felt at the entrance to the vagina (i.e. the vulvar vestibule) when pressure is applied to this area or during attempts at vaginal insertional activities (i.e. provoked).
  Interventions: Diagnostic Test: Corticomotor excitability to the pelvic floor muscles; Diagnostic Test: Pelvic floor muscle response to pressure applied at the vulvar vestibule; Diagnostic Test: Pressure pain threshold (PPS); Diagnostic Test: Temporal summation of pain; Diagnostic Test: Tonic, phasic and reflex activation of the pelvic floor muscles (PFMs)
- Provoked vestibulodynia (PVD) + Vaginismus (VAG): PVD is sometimes accompanied by intense, involuntary contraction of the PFMs3, termed vaginismus (VAG).
  Interventions: Diagnostic Test: Corticomotor excitability to the pelvic floor muscles; Diagnostic Test: Pelvic floor muscle response to pressure applied at the vulvar vestibule; Diagnostic Test: Pressure pain threshold (PPS); Diagnostic Test: Temporal summation of pain; Diagnostic Test: Tonic, phasic and reflex activation of the pelvic floor muscles (PFMs)
- Control: Participants matched by age (within 2 years), parity (parous vs nulliparous) and use of oral contraceptive medications (yes vs no) to women in the PVD group, with no signs and symptoms of PVD.
  Interventions: Diagnostic Test: Corticomotor excitability to the pelvic floor muscles; Diagnostic Test: Pelvic floor muscle response to pressure applied at the vulvar vestibule; Diagnostic Test: Pressure pain threshold (PPS); Diagnostic Test: Temporal summation of pain; Diagnostic Test: Tonic, phasic and reflex activation of the pelvic floor muscles (PFMs)

INTERVENTIONS:
Diagnostic Test: Corticomotor excitability to the pelvic floor muscles — Transcranial magenetic stimulation will be used to probe the excitability of cortical projections to the pelvic floor muscles. The outcomes of interest will include motor evoked potential amplitude and silent period.
Diagnostic Test: Pelvic floor muscle response to pressure applied at the vulvar vestibule — Electromyography will be used to determine whether the pelvic floor muscles (PFMs) respond to pressure applied to the vulvar vestibule as anticipatory (i.e. PFMs are active before the pressure is applied) and as behavioural (i.e. PFMs are active after the pressure is applied) responses. The amplitude of the EMG responses will also be recorded.
Diagnostic Test: Pressure pain threshold (PPS) — A custom vulvalgesiometer will be used to determine the mean pressure at which participants first report pain at the posterior vaginal fourchette.
Diagnostic Test: Temporal summation of pain — A custom vulvalgesiometer will be used to apply the same pressure (rated as 4/10 duiring PPS testing as described above) to the vulvar vestibule across 10 repetitions. The difference in pain rated on the tenth application and that rated on the first application will be the outcome.
Diagnostic Test: Tonic, phasic and reflex activation of the pelvic floor muscles (PFMs) — Electromyography will be used to measure the mean smoothed, rectified activation amplitude across 1 second of complete rest, across three maximal effort PFM contractions, and across three attempts at a bearing down maneuver.

SUMMARY:
Dyspareunia, or pain experienced by women during penetrative sexual activities, affects the psychological and sexual health of more than one in five Canadian women [1], yet its pathophysiology is poorly understood [2-4] and evidence for management approaches is limited.[5] It is thought that pelvic floor muscle (PFM) dysfunction is implicated in many forms of dyspareunia, while the nature and aetiology of this involvement remain largely unknown. The goal of this study is to understand if and how PFM dysfunction contributes to the pain experienced by women with provoked vestibulodynia (PVD), the most common cause of dyspareunia. This goal will be achieved through implementing an innovative and comprehensive approach to measuring the neuromuscular function of the PFMs. Understanding the pathophysiology of PVD is essential to the development of effective interventions to improve the health and quality of life of the many Canadian women who suffer from dyspareunia.

DETAILED DESCRIPTION:
Despite its high prevalence, little is known about the aetiology of dyspareunia. Dyspareunia is often sub-classified by the location (generalized vs a specific region) and by the stimulus that induces pain (provoked vs spontaneous). As such, PVD is characterized by severe sharp and/or burning pain felt at the entrance to the vagina (i.e. the vulvar vestibule) when pressure is applied to this area (i.e. provoked). [2] PVD is considered to be the most common cause of dyspareunia in pre-menopausal women, with a prevalence of about 12% of women, [1] while it remains underreported due to stigma embarrassment and shame. [6] Among women who seek intervention for PVD, involuntary PFM activation is thought to play a significant role in the onset and/or maintenance of pain. [7-15] Indeed, PVD is sometimes accompanied by intense, involuntary contraction of the PFMs [3], termed vaginismus (VAG). Yet it is not known whether PVD and VAG are distinct entities, or whether VAG exists along some continuum of PVD severity; [8,16] a matter of much debate in the literature.[17,19]

There is evidence to suggest that PFM dysfunction is a feature of PVD even in the absence of VAG.[7-15,20] When assessed through intravaginal palpation, women with PVD (without VAG) present with higher PFM tone (i.e., greater resistance to a passive manual stretch of the PFMs), difficulty relaxing their PFMs following a contraction, and lower PFM strength when compared to asymptomatic women.[7-9] Yet strength and tone graded by palpation are subjective, and studies were performed without assessor blinding. Some of these palpation findings have been corroborated using electromyography (EMG), including higher than normal tonic PFM activation,[14,21,22] poor ability to achieve a PFM contraction [10], impaired ability to relax the PFMs after activation [4], and/or poor ability to sustain a consistent activation level on voluntary PFM contraction,[10,15,23] yet the latter findings have been refuted by others.[9,20,24-26] While this more objective evidence exists, studies on PFM involvement in PVD using EMG have been small (n<12), have carried high risk of bias, [27] and authors have often failed to report whether women with PVD had concurrent VAG, perpetuating the lack of clarity around diagnosis.

Indeed, it is often difficult to determine on clinical examination whether or not VAG is present in women with PVD [3] and the new Diagnostic and Statistical Manual of Mental Disorders (DSM-5) omits any distinction between PVD and VAG, referring to both as genito pelvic pain penetration disorder (GPPPD17,21). Yet PFM involvement in PVD that is accompanied by VAG (PVD+VAG) may be distinct from PFM dysfunction in PVD with no concurrent VAG. [4,27-31] While trying to understand the nature of PFM involvement in PVD, it remains prudent to evaluate the PFMs while distinguishing between those with PVD+VAG and those with PVD alone.[19] This study will contribute to our knowledge of the nature of PFM involvement in PVD, and will inform on differences in PFM involvement between those with PVD alone and those with PVD+VAG.

Objectives and hypotheses: The overall goal of this project is to determine whether alterations in tonic, voluntary, reflex or behavioural responses of the superficial and/or the deep layer of the (PFMs) are implicated in PVD and/or PVD+VAG. There are four main aims with associated hypotheses:

Aim 1: To measure and compare pressure pain threshold (PPT), Temporal Summation (TS) at the vulvar vestibule, pain reported during the tampon test, and sexual function.

Hypothesis 1 (a): Compared to pain-free controls, women with PVD and PVD+VAG will demonstrate (a) greater self-reported pain during the tampon test. (b) lower PPT, (c) higher TS, and (d) lower sexual function.

Aim 2: To measure corticomotor excitability of projections to the PFMs through motor evoked potentials (MEPs) and cortically mediated silent periods (cSPs).

Hypothesis 2(a) Compared to pain-free controls, women with PVD and PVD+VAG will have larger MEPs and shorter cSPs in the bulbocavernosus, pubovisceral, and external anal sphincter muscles in response to transcranial magnetic stimulation (TMS) of the cortical area corresponding to the PFMs.

Hypothesis 2(b) Differences will be evident between women with PVD and PVD+VAG.

Aim 3: To measure the amplitude and timing of EMG responses to pressure applied to the vulvar vestibule and the posterior thigh Hypothesis 3 (a): Compared to pain-free controls, women with PVD and PVD+VAG will have higher incidences of anticipatory responses (ie. responses recorded before pressure is applied) recorded from the PFMs (bulbocavernosus, pubovisceral, external anal sphincter) and remote (uppper trapezius, hip adductor) muscles when standardized pressure stimuli are applied to the posterior vaginal fourchette regardless of the intensity of the pressure (low vs moderate).

Hypothesis 3 (b): Compared to pain-free controls, women with PVD and PVD+VAG will have higher muscle activation amplitude responses in the PFMs (bulbocavernosus, pubovisceral, external anal sphincter) and in more remote muscles (trapezius and hip adductor muscles) after standardized pressure stimuli (both low and moderate) are applied to the posterior vaginal fourchette.

Hypothesis 3 (c): Compared to pain-free controls, women with PVD and PVD+VAG will demonstrate larger responses in the PFMs (bulbocavernosus, pubovisceral, external anal sphincter) and in more remote muscles (trapezius or hip adductors) in response to pressure that is applied to the posterior thigh.

Aim 4: To measure the amplitude of PFM activation at rest (tonic), during maximum effort voluntary contraction of the PFMs and during a straining (Valsalva) maneuver Hypothesis 4: Compared to pain-free controls, women with PVD and PVD+VAG will demonstrate (a) higher tonic PFM activation, (b) more PFM activation during straining efforts (dyssynergia) and (c) lower PFM activation on maximum voluntary contraction.

Novelty and Contributions to the advancement of knowledge: Through this study, a comprehensive picture of neuromuscular impairments in the PFMs that are associated with PVD will be generated. Through Aim 1 it is expected to find in women with PVD and PVD+VAG, greater self reported pain during tampon test, lower pressure pain threshold, higher temporal summation and lower sexual function comparing with the control group. No study has investigated corticomotor excitability of projections to the PFMs through TMS. Through Aim 2 differences in corticomotor excitability to the PFMs, evidenced through higher amplitude MEPs and shorter duration cSPs are expected to be found, between women with and without PVD as well as differences in the extent of enhanced corticomotor excitability to the PFMs between PVD and PVD+VAG. Also no study has evaluated whether differences seen in tonic or phasic responses of the PFMs between women with PVD and controls are present because of or in anticipation of pain. Studies by Van Lunsen & Ramakers [32], Reissing et al. [8] and van der Velde & Everaerd [33] suggest that the PFMs respond to generalized anxiety and in response to watching sexually threatening scenes. It is quite possible, and even probable, that anxiety or fear of pain may influence study outcomes [4,34]. Through Aim 3, the timing and magnitude of PFM activation will be evaluated to determine whether responses occur in anticipation of (i.e. before) and/or in response to pressure stimuli delivered at the vulvar vestibule. The hypotheses under Aims 2 and 3 have never before been tested and doing so will have a significant impact on our understanding of the pathophysiology of PVD. Through Aim 4, it we expect to corroborate previous findings in the literature: that women with PVD and PVD+VAG will demonstrate higher tonic PFM activation and PFM dyssynergia during straining - both being functionally related to increased corticomotor excitability.

If women with PVD+VAG exhibit higher corticomotor excitability than women with PVD alone, this finding will be a major step toward understanding PVD and PVD+VAG as separate conditions, and will set the stage for improved diagnoses and targeted treatments such as repetitive TMS35 and neurotropic medications.[36] Further, interventions that have shown some evidence for effectiveness [37] including stretching, [9,38,39] acupuncture, [40] Botox injection, [41,42] and cognitive behavioural therapy [39] may be enhanced by combining them with new interventions that focus on corticomotor inhibition. The impact of any new as well as existing interventions on corticomotor excitability can, in turn, be evaluated using the innovative yet accessible assessment approaches developed through this work.

For descriptive purposes, five on-line questionnaires will be applied to assess sexual function [43,44], pain [45] pain catastrophising [46], depression/anxiety [47,48], and central sensitization [49].

Assessment will be scheduled within the week following the start of women's last menstrual cycle to account for cyclic variations in motor and sensory thresholds [50] , and at a time that is convenient.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women over the age of 18
* Biologically born female
* Signs and symptoms consistent with Provoked Vestibulodynia (PVD) alone or PVD+ Vaginismus (VAG) (i.e. evidence of a vaginal muscle spasm in response to palpation) or no history of pain during sexual activities or tampon insertion to serve as a comparison group
* Not currently pregnant, or pregnant in the past six months.

Exclusion Criteria:

* Neurological condition such as stroke, multiple sclerosis, spinal cord injury, epilepsy, or history of epilepsy in the family, etc
* Metal implants (cochlear, pacemaker, etc.)
* Tendency to faint
* in Peri- or post-menopause
* express high levels of anxiety about the assessment protocol

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Females with PVD alone or PVD+ VAG will be recruited at the vulvar pain clinic at The Ottawa Hospital and from local physiotherapy clinics that cater to females with pelvic floor dysfunction.
  Control participants will be recruited from the local community through advertisements, word of mouth and social media.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Motor evoked potential (MEP) peak to peak amplitude (µV) | 1 day
  Transcranial magnetic stimulation outcome (i.e. Motor evoked potential peak to peak amplitude - µV) will be determined for all participants and compared among groups.
  A Magstim® 200 system coupled with a double cone coil (96 mm loops, P/N 9902) [57] will be used to probe the corticospinal projections to PFMs. MEPs will be ensemble averaged to generate estimates of MEP peak to peak amplitude (µV).
Cortical silent period duration (ms) | 1 day
  Transcranial magnetic stimulation outcome (i.e. cortical silent period duration - ms) will be determined for all participants and compared among groups.
  A Magstim® 200 system coupled with a double cone coil (96 mm loops, P/N 9902) [57] will be used to probe the corticospinal projections to PFMs. MEP cortical silent period (cSP) will be measured from individual trials and then averaged.
Anticipatory responses (ms) | 1 day
  The proportion of women in each group who demonstrate anticipatory responses of the PFMs to impending pressure applied at the vulvar vestibule will be determined for each group. Participants will be deemed to have anticipatory responses if electromyographic signals recorded from the PFMs precede the application of pressure. A vulvalgesiometer [58] will be employed using a response-dependent methodology. [59,60] The vulvalgesiometer will be used to apply low (25 g) and moderate (232 g) pressures to the posterior vaginal fourchette or to the posterior thigh, the moderate value having been generated through the team's previous research. [9]
Behavioural responses (µV) | 1 day
  The proportion of women in each group who demonstrate behavioral responses of the PFMs to pressure applied at the vulvar vestibule will be determined for each group. Participants will be deemed to have behavioural if the activation of the PFMs (or other muscles) occurs after the pressure is applied. A vulvalgesiometer [58] will be employed using a response-dependent methodology. [59,60] The vulvalgesiometer will be used to apply low (25 g) and moderate (232 g) pressures to the posterior vaginal fourchette or to the posterior thigh, the moderate value having been generated through the team's previous research. [9]
Tonic, phasic and reflex activation of the pelvic floor muscles | 1 day
  Surface Electromyography (EMG) recorded using differential suction electrodes (DSEs, developed by Dr. McLean) [54-56] will be used to measure tonic, voluntary and reflex activation of the superficial and deep PFMs. Smoothed peak EMG amplitudes (µV) will be computed as outcomes while women keep their PFMs as relaxed as possible (tonic), contract as strongly as possible (phasic) and perform a straining maneuver (reflex activation).

SECONDARY OUTCOMES:
Tampon test | 1 day
  Women will be instructed to insert and then remove the tampon and they will be instructed to record the degree of pain during the entire insertion/ removal experience on a 0-10 pain numeric rating scale, with 0 meaning no pain, and 10 meaning the worst possible pain.
Pressure pain threshold (PPT) | 1 day
  The pressure at which women report pain on pressure applied through a cotton swab to the region of the posterior vaginal fourchette.
  Pressure pain threshold (PPT) will be determined using a custom vulvalgesiometer. PPT will be defined as the average pressure at which women first report pain when the cotton swab tip of the vulvalgesiometer is applied at 6 o' clock of the vaginal introitus [51].
Temporal summation (TS) of pain | 1 day
  The difference in pain rating (scale 1-10) between the tenth and first application of a pressure applied to the posterior vaginal fourchette through a custom vulvalgesiometer.
  The PPT determined at the 6-o-clock position, will be applied ten times at a rate of approximately one per second at the 6 o'clock location on the vestibule. Participants will rate their pain level on the initial and final application of this pressure using a Numeric Rating Scale (0-10). TS will be defined as the difference in pain rating between the final and first application of the pressure [52,53]

OTHER OUTCOMES:
Female sexual function index (FSFI) | 1 day
  This is a 19-item validated questionnaire [43,44] for assessing the key dimension of sexual function in women, considered a gold standard for evaluation of sexual function. It assesses six domains: desire, arousal , lubrification, orgasm, satisfaction, and pain. All scores are totaled for a maximum of 36. Higher scores represents better sexual function. A score ≤26.55 has been set as a cutoff to identify those at risk for sexual dysfunction.
McGill Pain Questionnaire | 1 day
  This questionnaire consists primarily of 3 major classes of word descriptors - sensory, affective and evaluative - that are used by patients to specify subjective pain experience. It also contains an intensity scale and other items to determine the properties of pain experience. This questionnaire is composed of 78 words. Respondents choose those that best describe their experience of pain. Scores are tabulated by summing values associated with each word; scores range from 0 (no pain) to 78 (severe pain). Quantitative differences in pain may be reflected in respondents word choice.
Pain catastrophizing scale | 1 day
  The Pain Catastrophizing Scale is a reliable and valid measure of catastrophizing. The scores from this questionnaire is predictors of intensity of physical and emotional distress.
  It is a self-report measure, consisting of 13 items scored from 0 to 4, resulting in a total possible score of 52. The higher the score, the more catastrophizing thoughts are present
Depression Anxiety Stress Scale (DASS) | 1 day
  This is a 42-item self report instrument designed to measure the three related negative emotional states of depression, anxiety and tension/stress [47,48]. Each one contains 14 items, divided into subscales of 2-5 items with similar content. The DASS have been shown to have high internal consistency and to yield meaningful discriminations in a variety of settings.
  A higher score on the DASS indicates greater severity or frequency of these negative emotional symptoms. The maximum score is 126.
Central sensitization inventory | 1 day
  The Central Sensitisation Inventory (CSI) [49], is a self-report outcome measure designed to identify patients who have symptoms that may be related to central sensitisation (CS) or central sensitivity syndromes (CSS). Part A includes 25 questions related to common CSS symptoms.
  Part B determines if the patient has been diagnosed with certain CSS disorders or related disorders, such as anxiety and depression. CSI severity levels have been established for part A: subclinical = 0 to 29; mild = 30 to 39; moderate = 40 to 49; severe = 50 to 59; and extreme = 60 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Linda McLean, Principal Investigator — University of Ottawa
Locations (1):
- Flavia Antonio, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Spreadsheets will be provided by email upon request and based on the planned use of the data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available for 10 years after the publication of the study results.
Access Criteria: Planned use of data for systematic review.

REFERENCES:
- [Background] Harlow BL, Stewart EG. A population-based assessment of chronic unexplained vulvar pain: have we underestimated the prevalence of vulvodynia? J Am Med Womens Assoc (1972). 2003 Spring;58(2):82-8. PMID 12744420
- [Background] Bergeron S, Binik YM, Khalife S, Pagidas K, Glazer HI. Vulvar vestibulitis syndrome: reliability of diagnosis and evaluation of current diagnostic criteria. Obstet Gynecol. 2001 Jul;98(1):45-51. doi: 10.1016/s0029-7844(01)01389-8. PMID 11430955
- [Background] de Kruiff ME, ter Kuile MM, Weijenborg PT, van Lankveld JJ. Vaginismus and dyspareunia: is there a difference in clinical presentation? J Psychosom Obstet Gynaecol. 2000 Sep;21(3):149-55. doi: 10.3109/01674820009075622. PMID 11076336
- [Background] Lahaie MA, Amsel R, Khalife S, Boyer S, Faaborg-Andersen M, Binik YM. Can Fear, Pain, and Muscle Tension Discriminate Vaginismus from Dyspareunia/Provoked Vestibulodynia? Implications for the New DSM-5 Diagnosis of Genito-Pelvic Pain/Penetration Disorder. Arch Sex Behav. 2015 Aug;44(6):1537-50. doi: 10.1007/s10508-014-0430-z. Epub 2014 Nov 15. PMID 25398588
- [Background] Andrews JC. Vulvodynia interventions--systematic review and evidence grading. Obstet Gynecol Surv. 2011 May;66(5):299-315. doi: 10.1097/OGX.0b013e3182277fb7. PMID 21794194
- [Background] Donaldson RL, Meana M. Early dyspareunia experience in young women: confusion, consequences, and help-seeking barriers. J Sex Med. 2011 Mar;8(3):814-23. doi: 10.1111/j.1743-6109.2010.02150.x. Epub 2010 Dec 8. PMID 21143423
- [Background] Reissing ED, Brown C, Lord MJ, Binik YM, Khalife S. Pelvic floor muscle functioning in women with vulvar vestibulitis syndrome. J Psychosom Obstet Gynaecol. 2005 Jun;26(2):107-13. doi: 10.1080/01443610400023106. PMID 16050536
- [Background] Reissing ED, Binik YM, Khalife S, Cohen D, Amsel R. Vaginal spasm, pain, and behavior: an empirical investigation of the diagnosis of vaginismus. Arch Sex Behav. 2004 Feb;33(1):5-17. doi: 10.1023/B:ASEB.0000007458.32852.c8. PMID 14739686
- [Background] Gentilcore-Saulnier E, McLean L, Goldfinger C, Pukall CF, Chamberlain S. Pelvic floor muscle assessment outcomes in women with and without provoked vestibulodynia and the impact of a physical therapy program. J Sex Med. 2010 Feb;7(2 Pt 2):1003-22. doi: 10.1111/j.1743-6109.2009.01642.x. Epub 2010 Jan 6. PMID 20059663
- [Background] Glazer HI, Rodke G, Swencionis C, Hertz R, Young AW. Treatment of vulvar vestibulitis syndrome with electromyographic biofeedback of pelvic floor musculature. J Reprod Med. 1995 Apr;40(4):283-90. PMID 7623358
- [Background] Morin M, Bergeron S, Khalife S, Mayrand MH, Binik YM. Morphometry of the pelvic floor muscles in women with and without provoked vestibulodynia using 4D ultrasound. J Sex Med. 2014 Mar;11(3):776-85. doi: 10.1111/jsm.12367. Epub 2013 Nov 6. PMID 24344835
- [Background] 12. Morin M, Bergeron S, Khalife S, Binik I, Ouellet S. Dynamometric assessment of the pelvic floor muscle function in women with and without provoked vestibulodynia. Int Urogynecol J 2010: 21: S336-S37.
- [Background] McKay E, Kaufman RH, Doctor U, Berkova Z, Glazer H, Redko V. Treating vulvar vestibulitis with electromyographic biofeedback of pelvic floor musculature. J Reprod Med. 2001 Apr;46(4):337-42. PMID 11354833
- [Background] Frasson E, Graziottin A, Priori A, Dall'ora E, Didone G, Garbin EL, Vicentini S, Bertolasi L. Central nervous system abnormalities in vaginismus. Clin Neurophysiol. 2009 Jan;120(1):117-22. doi: 10.1016/j.clinph.2008.10.156. Epub 2008 Dec 13. PMID 19071060
- [Background] White G, Jantos M, Glazer H. Establishing the diagnosis of vulvar vestibulitis. J Reprod Med. 1997 Mar;42(3):157-60. PMID 9109083
- [Background] Steege JF, Zolnoun DA. Evaluation and treatment of dyspareunia. Obstet Gynecol. 2009 May;113(5):1124-1136. doi: 10.1097/AOG.0b013e3181a1ba2a. PMID 19384129
- [Background] Binik YM. The DSM diagnostic criteria for dyspareunia. Arch Sex Behav. 2010 Apr;39(2):292-303. doi: 10.1007/s10508-009-9563-x. PMID 19830537
- [Background] Binik YM. The DSM diagnostic criteria for vaginismus. Arch Sex Behav. 2010 Apr;39(2):278-91. doi: 10.1007/s10508-009-9560-0. PMID 19851855
- [Background] Reissing ED, Borg C, Spoelstra SK, Ter Kuile MM, Both S, de Jong PJ, van Lankveld JJ, Melles RJ, Weijenborg PT, Weijmar Schultz WC. "Throwing the baby out with the bathwater": the demise of vaginismus in favor of genito-pelvic pain/penetration disorder. Arch Sex Behav. 2014 Oct;43(7):1209-13. doi: 10.1007/s10508-014-0322-2. No abstract available. PMID 25024064
- [Background] Engman M, Lindehammar H, Wijma B. Surface electromyography diagnostics in women with partial vaginismus with or without vulvar vestibulitis and in asymptomatic women. J Psychosom Obstet Gynaecol. 2004 Sep-Dec;25(3-4):281-94. doi: 10.1080/01674820400017921. PMID 15715027
- [Background] Shafik A, El-Sibai O. Study of the pelvic floor muscles in vaginismus: a concept of pathogenesis. Eur J Obstet Gynecol Reprod Biol. 2002 Oct 10;105(1):67-70. doi: 10.1016/s0301-2115(02)00115-x. PMID 12270568
- [Background] 22. Gammoudi N, Affes Z, Mellouli S, Radhouane K, Dogui M. The diagnosis value of needle electrode electromyography in vaginismus. Sexologies 2016: 25:e57-60. doi:10.1016/j.sexol.2016.04.005.
- [Background] Glazer HI, Jantos M, Hartmann EH, Swencionis C. Electromyographic comparisons of the pelvic floor in women with dysesthetic vulvodynia and asymptomatic women. J Reprod Med. 1998 Nov;43(11):959-62. PMID 9839264
- [Background] Naess I, Bo K. Pelvic floor muscle function in women with provoked vestibulodynia and asymptomatic controls. Int Urogynecol J. 2015 Oct;26(10):1467-73. doi: 10.1007/s00192-015-2660-6. Epub 2015 Mar 4. PMID 25735988
- [Background] McLean L, Thibault-Gagnon S, Brooks K, Goldfinger C, Pukall C, Chamberlain S. Differences in Pelvic Morphology Between Women With and Without Provoked Vestibulodynia. J Sex Med. 2016 Jun;13(6):963-71. doi: 10.1016/j.jsxm.2016.04.066. PMID 27215690
- [Background] Thibault-Gagnon S, McLean L, Goldfinger C, Pukall C, Chamberlain S. Differences in the Biometry of the Levator Hiatus at Rest, During Contraction, and During Valsalva Maneuver Between Women With and Without Provoked Vestibulodynia Assessed by Transperineal Ultrasound Imaging. J Sex Med. 2016 Feb;13(2):243-52. doi: 10.1016/j.jsxm.2015.12.009. Epub 2016 Jan 21. PMID 26805942
- [Background] 27. Gentilcore-Saulnier E, Auchincloss C, McLean L. Electromyography. In: Padoa A, Rosenbaum TY, editors. The Overactive Pelvic Floor. 1st ed., Springer International Publishing; 2016, p. 175-203. doi:10.1007/978-3-319-22150-2_12.
- [Background] McLean L, Brooks K. What Does Electromyography Tell Us About Dyspareunia? Sex Med Rev. 2017 Jul;5(3):282-294. doi: 10.1016/j.sxmr.2017.02.001. Epub 2017 Mar 18. PMID 28330675
- [Background] Maseroli E, Scavello I, Cipriani S, Palma M, Fambrini M, Corona G, Mannucci E, Maggi M, Vignozzi L. Psychobiological Correlates of Vaginismus: An Exploratory Analysis. J Sex Med. 2017 Nov;14(11):1392-1402. doi: 10.1016/j.jsxm.2017.09.015. PMID 29110807
- [Background] Ciocca G, Limoncin E, Di Tommaso S, Gravina GL, Di Sante S, Carosa E, Tullii A, Marcozzi A, Lenzi A, Jannini EA. Alexithymia and vaginismus: a preliminary correlation perspective. Int J Impot Res. 2013 May;25(3):113-6. doi: 10.1038/ijir.2013.5. Epub 2013 Mar 7. PMID 23466663
- [Background] Melles RJ, ter Kuile MM, Dewitte M, van Lankveld JJ, Brauer M, de Jong PJ. Automatic and deliberate affective associations with sexual stimuli in women with lifelong vaginismus before and after therapist-aided exposure treatment. J Sex Med. 2014 Mar;11(3):786-99. doi: 10.1111/jsm.12360. Epub 2013 Oct 25. PMID 24165436
- [Background] 32. Van Lunsen RHW, Ramakers MJ. The hyperactive pelvic floor syndrome (HPFS): psychosomatic and psycho-sexual aspects of hyperactive pelvic floor disorders with co-morbidity of uro-gynaecological, gastrointestinal and sexual symptomatology. Acta Endoscopica 2002: 32:275-85. doi:10.1007/BF03020230.
- [Background] van der Velde J, Everaerd W. The relationship between involuntary pelvic floor muscle activity, muscle awareness and experienced threat in women with and without vaginismus. Behav Res Ther. 2001 Apr;39(4):395-408. doi: 10.1016/s0005-7967(00)00007-3. PMID 11280339
- [Background] Vandyken C, Hilton S. Physical Therapy in the Treatment of Central Pain Mechanisms for Female Sexual Pain. Sex Med Rev. 2017 Jan;5(1):20-30. doi: 10.1016/j.sxmr.2016.06.004. Epub 2016 Aug 3. PMID 27498209
- [Background] Naro A, Milardi D, Russo M, Terranova C, Rizzo V, Cacciola A, Marino S, Calabro RS, Quartarone A. Non-invasive Brain Stimulation, a Tool to Revert Maladaptive Plasticity in Neuropathic Pain. Front Hum Neurosci. 2016 Jul 27;10:376. doi: 10.3389/fnhum.2016.00376. eCollection 2016. PMID 27512368
- [Background] Fassoulaki A, Sarantopoulos C, Melemeni A, Hogan Q. EMLA reduces acute and chronic pain after breast surgery for cancer. Reg Anesth Pain Med. 2000 Jul-Aug;25(4):350-5. doi: 10.1053/rapm.2000.7812. PMID 10925929
- [Background] Morin M, Carroll MS, Bergeron S. Systematic Review of the Effectiveness of Physical Therapy Modalities in Women With Provoked Vestibulodynia. Sex Med Rev. 2017 Jul;5(3):295-322. doi: 10.1016/j.sxmr.2017.02.003. Epub 2017 Mar 28. PMID 28363763
- [Background] Goldfinger C, Pukall CF, Gentilcore-Saulnier E, McLean L, Chamberlain S. A prospective study of pelvic floor physical therapy: pain and psychosexual outcomes in provoked vestibulodynia. J Sex Med. 2009 Jul;6(7):1955-68. doi: 10.1111/j.1743-6109.2009.01304.x. Epub 2009 Apr 28. PMID 19453890
- [Background] Goldfinger C, Pukall CF, Thibault-Gagnon S, McLean L, Chamberlain S. Effectiveness of Cognitive-Behavioral Therapy and Physical Therapy for Provoked Vestibulodynia: A Randomized Pilot Study. J Sex Med. 2016 Jan;13(1):88-94. doi: 10.1016/j.jsxm.2015.12.003. PMID 26755091
- [Background] Schlaeger JM, Xu N, Mejta CL, Park CG, Wilkie DJ. Acupuncture for the treatment of vulvodynia: a randomized wait-list controlled pilot study. J Sex Med. 2015 Apr;12(4):1019-27. doi: 10.1111/jsm.12830. Epub 2015 Jan 30. PMID 25639289
- [Background] Pelletier F, Parratte B, Penz S, Moreno JP, Aubin F, Humbert P. Efficacy of high doses of botulinum toxin A for treating provoked vestibulodynia. Br J Dermatol. 2011 Mar;164(3):617-22. doi: 10.1111/j.1365-2133.2011.10235.x. PMID 21275944
- [Background] Bertolasi L, Frasson E, Cappelletti JY, Vicentini S, Bordignon M, Graziottin A. Botulinum neurotoxin type A injections for vaginismus secondary to vulvar vestibulitis syndrome. Obstet Gynecol. 2009 Nov;114(5):1008-1016. doi: 10.1097/AOG.0b013e3181bb0dbb. PMID 20168100
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Background] Meyer-Bahlburg HF, Dolezal C. The female sexual function index: a methodological critique and suggestions for improvement. J Sex Marital Ther. 2007 May-Jun;33(3):217-24. doi: 10.1080/00926230701267852. PMID 17454519
- [Background] Melzack R. The McGill Pain Questionnaire: major properties and scoring methods. Pain. 1975 Sep;1(3):277-299. doi: 10.1016/0304-3959(75)90044-5. PMID 1235985
- [Background] 46. Sullivan, M. J. L., Bishop, S. R., &Pivik, J. The Pain Catastrophizing Scale: Development and validation. Psychological Assessment 1995; 7, 524-532.
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] 48. Lovibond, S.H.; Lovibond, P.F.
- [Background] Mayer TG, Neblett R, Cohen H, Howard KJ, Choi YH, Williams MJ, Perez Y, Gatchel RJ. The development and psychometric validation of the central sensitization inventory. Pain Pract. 2012 Apr;12(4):276-85. doi: 10.1111/j.1533-2500.2011.00493.x. Epub 2011 Sep 27. PMID 21951710
- [Background] Barbosa Mde B, Guirro EC, Nunes FR. Evaluation of sensitivity, motor and pain thresholds across the menstrual cycle through medium-frequency transcutaneous electrical nerve stimulation. Clinics (Sao Paulo). 2013 Jul;68(7):901-8. doi: 10.6061/clinics/2013(07)03. PMID 23917651
- [Background] Pukall CF, Young RA, Roberts MJ, Sutton KS, Smith KB. The vulvalgesiometer as a device to measure genital pressure-pain threshold. Physiol Meas. 2007 Dec;28(12):1543-50. doi: 10.1088/0967-3334/28/12/008. Epub 2007 Dec 3. PMID 18057518
- [Background] Petersen KK, Arendt-Nielsen L, Simonsen O, Wilder-Smith O, Laursen MB. Presurgical assessment of temporal summation of pain predicts the development of chronic postoperative pain 12 months after total knee replacement. Pain. 2015 Jan;156(1):55-61. doi: 10.1016/j.pain.0000000000000022. PMID 25599301
- [Background] Weissman-Fogel I, Granovsky Y, Crispel Y, Ben-Nun A, Best LA, Yarnitsky D, Granot M. Enhanced presurgical pain temporal summation response predicts post-thoracotomy pain intensity during the acute postoperative phase. J Pain. 2009 Jun;10(6):628-36. doi: 10.1016/j.jpain.2008.12.009. Epub 2009 Apr 23. PMID 19398382
- [Background] Keshwani N, McLean L. Development of a differential suction electrode for improved intravaginal recordings of pelvic floor muscle activity: reliability and motion artifact assessment. Neurourol Urodyn. 2012 Nov;31(8):1272-8. doi: 10.1002/nau.22253. Epub 2012 Jun 5. PMID 22674421
- [Background] Keshwani N, McLean L. A differential suction electrode for recording electromyographic activity from the pelvic floor muscles: crosstalk evaluation. J Electromyogr Kinesiol. 2013 Apr;23(2):311-8. doi: 10.1016/j.jelekin.2012.10.016. Epub 2012 Dec 5. PMID 23218961
- [Background] Keshwani N, McLean L. State of the art review: Intravaginal probes for recording electromyography from the pelvic floor muscles. Neurourol Urodyn. 2015 Feb;34(2):104-12. doi: 10.1002/nau.22529. Epub 2013 Nov 21. PMID 24264797
- [Background] 57. Hovey, C., & Jalinous, R. The guide to magnetic stimulation. Magstim Company Ltd July. 2006.
- [Background] 58. Pukall CF, Dawson S, Young R, Yessick L, Goldfinger C, Sutton KS, Dargie EE, Chamberlain SM.Journal of Sexual Medicine. (Submitted November 2017).
- [Background] Moseley GL, Arntz A. The context of a noxious stimulus affects the pain it evokes. Pain. 2007 Dec 15;133(1-3):64-71. doi: 10.1016/j.pain.2007.03.002. Epub 2007 Apr 20. PMID 17449180
- [Background] Tracy LM, Gibson SJ, Georgiou-Karistianis N, Giummarra MJ. Effects of explicit cueing and ambiguity on the anticipation and experience of a painful thermal stimulus. PLoS One. 2017 Aug 23;12(8):e0183650. doi: 10.1371/journal.pone.0183650. eCollection 2017. PMID 28832636